CLINICAL TRIAL: NCT02771314
Title: A Longitudinal Study Evaluating Molecular Changes Associated With Resistance to First and Third (AZD9291) Generation EGFR TKIs in Patients With EGFR Mutant NSCLC Using "Liquid Biopsy"
Brief Title: Liquid Biopsy as a Tool to Evaluate Resistance to First and Third (AZD9291) (EGFR) (TKIs) in (EGFR) Mutant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5160C00030
Record Dates: First submitted 2016-04-12; First posted 2016-05-13 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; AZD9291; >= 2nd line; liquid biopsy; EGFR TKIs; EGFR mutant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 (Experimental): AZD9291
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — AZD9291, 80 mg (tablets) once daily, administered orally in the fasted state
  Other Names: Tagrisso; Osimertinib

SUMMARY:
Based on the possibilities that both plasma and circulating tumor cells (CTCs) (the "liquid biopsy") may offer, we consider that it could be feasible to longitudinally monitor the genetic evolution and the biologic characteristics of CTCs, by using Circulating tumor DNA (ctDNA) and CTCs as a source of biologic material. This approach could provide information regarding the genetic/molecular changes associated with primary and acquired resistance to AZD9291 and, thus, to facilitate to more appropriately adapt the tailored treatment in this particular group of NSCLC patients. It has been recently reported that the detection of resistant clones, based on the tumor-associated genetic aberrations in the blood, can identify treatment resistance up to 10 months earlier than the radiological methods providing, thus, the potential for an early switch to a non cross-resistant therapy in order to improve patients' outcome.

DETAILED DESCRIPTION:
Lung cancer is among the most common tumor types representing 13% of the newly diagnosed cancers worldwide. Both the absolute and relative frequency of lung cancer has risen dramatically. Unfortunately, lung cancer remains by far the leading cause of cancer-related deaths, accounting for 18% of the total number of deaths. Non Small Lung Cancer (NSCLC) accounts for 85% of all cases of lung cancer and is further classified in several subtypes based on various molecular and histological features.

The initial dose of 80 mg AZD9291 administered once daily orally in the fasted state can be reduced to 40 mg AZD9291 once daily under circumstances

Single arm, open-label, phase II, multicenter study. NSCLC patients with activating EGFR mutations, who are under front line treatment with first generation EGFR TKIs according to the physicians' choice and present disease progression, will be treated with single agent AZD9291. The patients will be followed every 3 months for the detection of mutations (T790M), (C797S), (L858R), del 19 EGFR mutations as well as the mutations [(KRAS)/(NRAS), (BRAF), (PI3K)] in the serum/plasma, the determination of the serum levels of Hepatocyte Growth Factor (HGF), the presence of T790M (+) and C797S(+) CTCs as well as the molecular (c-MET) and (HER2 amplification) and phenotypic characterization of CTCs using the filtration platform (ISET). The elimination or the emergence of each of these circulating tumor biomarkers will be correlated with patients' clinical outcome [objective response to treatment (ORR), (PFS) and (OS)].

There is no specific control group in this study. Biomarkers profile at baseline will be used as internal control for each patient to monitor changes throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Both sexes
3. Histologically or cytologically documented NSCLC
4. Stage 3b (IIIb) not amenable to radical therapy or stage IV
5. Presence of EGFR activating mutations (exon 19 deletion or L858R in exon 21)
6. First or second line treatment with EGFR TKIs
7. Performance status (ECOG): 0-1
8. Measurable or evaluable disease
9. Adequate organ function tests (Hb>=10g/dL, white blood cell (WBC) >=3.0 x 10^9/L, neutrophils count >=1.5 x 10^9/L, platelets≥100 x 10^9/L, Creatinine clearance >=50 mL/min, Total bilirubin=<1.5 X UNL, aspartate aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline phosphatase (ALP) =<2.5 x UNL)
10. Normal QT interval in ECG
11. Central nervous system (CNS) metastases are allowed provided that they have been irradiated and the patient is clinically stable
12. Women of child bearing potential and all men will be required to use adequate contraceptive measures
13. Life expectancy of at least 3 months
14. Written informed consent

Exclusion Criteria:

1. History of serious drug allergy
2. Refractory nausea, vomiting and chronic gastrointestinal diseases
3. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
4. Severe or uncontrolled systemic liver disease, including those with known hepatitis B, hepatitis C, and Human Immunodeficiency virus (HIV) infection
5. Interstitial lung disease or pulmonary fibrosis
6. Pregnancy, lactation or other concomitant serious medical condition
7. Other concurrent active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of resistance to first and third (AZD9291) generation EGFR TKIs, explored by studying baseline serial serum or plasma DNA specimens and baseline Circulating Tumor Cells (CTCs) | Up to 2.5 years

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2.5 years
Overall Survival | Up to 2.5 years
Response rate, assessed using RECIST 1.1 | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Kotsakis, PhD, Principal Investigator — Hellenic Oncology Research Group
Locations (13):
- Greece (13):
  - University Hospital of Heraklion Crete, Heraklion, Crete
  - 251 Air Forces Military Hospital of Athens, Athens
  - Anticancer Hospital of Athens "Agios Savvas", Athens
  - Athens Hospital "Mitera" Hygia Polis, Athens
  - General Hospital of Athens "Aretaieio", Athens
  - General Hospital of Athens "Evangelismos", Athens
  - General Oncology Hospital of Athens "Ag. Anargiroi", Athens
  - IASO General Hospital, Athens
  - Universtiy Hospital of Athens "Attikon", Athens
  - University Hospital of Patra-Rio, Rio
  - Diabalkaniko General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thesaloniki "G. Papanikolaou", Thessaloniki
  - Thessaloniki Bioclinic, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided